CLINICAL TRIAL: NCT05127109
Title: The PASTDUe Nutrition EcoSystem Pathway In Acute Care Abdominal Surgery and Trauma to Decrease Underfeeding and Complications
Brief Title: The PASTDUe Nutrition Ecosystem Project (PASTDUe)
Acronym: PASTDUe
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00107553
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Diet, Healthy; Food; Nutrition; Intensive Care; Abdominal Trauma; Surgery; Intra-abdominal Infection; Sepsis; Ischemic Bowel; Vascular; Penetrating Abdominal Trauma; Enteral Feeding; Oral
MeSH Terms: conditions — Abdominal Injuries; Intraabdominal Infections; Sepsis

STUDY DESIGN:
Intervention Model Description: Utilization of structured nutrition delivery pathway on 300 adult abdominal trauma and surgery patients admitted to a Duke University Medical Center (DUMC) intensive care unit (ICU) from surgical intervention to hospital discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Nutrition Ecosystem pathway (Experimental): 1. parenteral nutrition initiated within 72 hours of operative intervention
  2. metabolic cart assessments to determine resting energy expenditure (REE) and guide registered dietitians (RDs)
  3. expedited delivery of oral nutrition supplements and
  4. a team-based approach on proper documentation of nutrition delivery and intake.
  Interventions: Combination Product: Nutrition Ecosystem pathway
- Comparator (Other): 300 historical matched control subjects not having received TPN in the first 7 hospital days will be enrolled from Duke Electronic Health Record between January 2018 and June 2020.
  Interventions: Other: Comparator

INTERVENTIONS:
Combination Product: Nutrition Ecosystem pathway — 1. parenteral nutrition initiated within 72 hours of operative intervention
     * Provided as clinically appropriate: Ensure Enlive, Ensure High-Protein, Nepro with Carb-Steady/ProSource Gelatein Plus, and/or ProSource Gelatein Plus
  2. metabolic cart assessments to determine resting energy expenditure (REE) and guide registered dietitians (RDs)
     * Q-NRG Metabolic Cart (Indirect Calorimeter) and Quark RMR Metabolic Cart (Indirect Calorimeter)
     * BWA 2.0 Advanced Bioelectric Impedance Spectroscopy (BIS)
     * Philips Lumify L12-4 broadband linear array transducer ultrasound
  3. expedited delivery of oral nutrition supplements and
  4. a team-based approach on proper documentation of nutrition delivery and intake
  Arms: Nutrition Ecosystem pathway
Other: Comparator — retrospective cohort of 300 historical matched control subjects
  Arms: Comparator

SUMMARY:
This is a research study to determine if a particular method of providing nutrition improves the clinical outcomes of patients in the intensive care unit (ICU) who have undergone abdominal surgery and would require nutrition delivered via the bloodstream (called total parenteral nutrition or TPN). The nutrition method we are testing is a structured nutrition delivery plan that involves tube feeding, oral nutrition supplements, and the use of a device (called an indirect calorimeter or IC) to measure calorie needs. This study will also use two devices to measure fat and muscle mass to examine changes during hospitalization. Subjects will be followed throughout hospitalization where nutrition status and fat and muscle mass will be closely monitored.

Study activities will begin within 72 hours of a patient's abdominal surgery. TPN (total parenteral nutrition, a method of feeding that bypasses the usual process of eating and digestion) will be started, a non-invasive method of assessing calorie needs (indirect calorimetry (IC)) will be started, a urine sample will be collected to help assist in protein needs, and fat/muscle mass will be measured using bioelectrical impedance analysis (BIA), and an ultrasound. This is a minimal risk study and all products/devices used are non-invasive and FDA-approved. Indirect calorimetry and urine sample collection will be conducted every 3 days during the stay in the Intensive Care Unit - ICU, then every 5 days until hospital discharge. BIA and muscle ultrasound will be conducted every 7 days during ICU stay, then every 14 days until hospital discharge.

DETAILED DESCRIPTION:
The purpose of this prospective trial is to study the impact of the utilization of structured nutrition delivery pathway on 300 adult abdominal trauma and surgery patients admitted to a Duke University Medical Center (DUMC) intensive care unit (ICU) through a structured nutrition delivery pathway from surgical intervention to hospital discharge. Objectives include evaluating the impact of a structured nutrition delivery pathway on 1) nosocomial infectious complications as defined by CDC guidelines after 7 days of ICU admission and 2) protein-calorie malnutrition, ventilator use, hospital disposition, hospital and ICU length of stay, ED/hospital utilization, total parenteral nutrition (TPN)-related complications, 1-year mortality, and hospital charges. Patient outcomes will be compared to a retrospective cohort of 300 historical matched control subjects.

The study intervention, a structured nutrition delivery pathway called the Nutrition Ecosystem pathway consists of the following collaborative parts to optimize nutrition intake and delivery within this patient population: 1) parenteral nutrition initiated within 72 hours of operative intervention 2) metabolic cart assessments to determine resting energy expenditure (REE) and guide registered dietitians (RDs) 3) expedited delivery of oral nutrition supplements and 4) a team-based approach on proper documentation of nutrition delivery and intake. The population group will consist of 300 surgical patients admitted to a DUMC ICU following emergent/urgent major abdominal surgery secondary to abdominal trauma, intra-abdominal sepsis, ischemic bowel/vascular emergencies, or penetrating trauma and are not expected to receive enteral or oral nutrition for at least 72 hours. 300 historical matched control subjects not having received TPN in the first 7 hospital days will be enrolled from Duke Electronic Health Record between January 2018 and June 2020.

This study poses minimal risks to patients as the study activities match the current standard of care medical treatment such as nutrition delivery via TPN. Patients will benefit from metabolic and physiologic assessments, closer monitoring, and interdisciplinary support for nutrition optimization from nurses, dietitians, and providers throughout their hospitalization. Given patients' energy expenditure will be routinely measured by indirect calorimetry via a metabolic cart, a greater accuracy in caloric requirements will help achieve precision and goal nutrition for all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. ICU admission with major abdominal trauma, intra-abdominal sepsis, ischemic bowel/vascular emergencies, or penetrating trauma
3. Not expected to receive oral or enteral nutrition for > 72 hours
4. Primary team approval of PN

4. < 72 hours post-operative intervention

Exclusion Criteria:

1. Expected death or withdrawal of life-sustaining treatment within the first 72 hours of ICU admission
2. Patients admitted with

   * Diabetic ketoacidosis or non-ketotic hyperosmolar coma
   * MELD > 20 or acute fulminant hepatic failure
3. Patients allergic to any component of parenteral nutrition or lipid solution
4. Pregnant or breastfeeding patients
5. Incarcerated or prisoner prior to admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of nosocomial infection complications as measured by medical record review | From TPN initiation, daily until hospital discharge (up to 8 months)
ICU length of stay in days measured by medical record review | From TPN initiation, daily until hospital discharge (up to 8 months)

SECONDARY OUTCOMES:
Incidence of protein-calorie malnutrition measured using AND/ASPEN-defined malnutrition criteria | Measured daily from hospital admission to hospital discharge (up to 8 months)
Number of days patient is on ventilator measured by medical record review | Measured daily from hospital admission up to hospital discharge (up to 8 months)
Number of patients discharged home measured by medical record review/patient report | Recorded at hospital discharge (up to 8 months)]
Number of patients discharged to rehabilitation center measured by medical record review/patient report | Recorded at hospital discharge (up to 8 months)]
Number of patients discharged to nursing home measured by medical record review/patient report | Recorded at hospital discharge (up to 8 months)]
ICU length of stay in days measured by medical record review | Measured from ICU admission to ICU discharge (up to 8 months)
Length of hospital stay in days as measured by medical record review | Measured from hospital admission to hospital discharge (up to 8 months)
Incidence of ED/hospital utilization as measured by medical record review/patient report | Measured from hospital discharge to 1-year post-hospital discharge]
Number of TPN-related complications as measured by medical record review/patient report | Measured from TPN initiation until completion of TPN course/treatment (up to 8 months)
Number of the different types of TPN-related complications as measured by medical record review/patient report | Measured from TPN initiation until completion of TPN course/treatment(up to 8 months)
Number of deaths in 1-year as measured by medical record review/Legally Authorized Representative report | Measured from hospital discharge to 1-year post-hospital discharge]

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wischmeyer, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No